CLINICAL TRIAL: NCT02096627
Title: Comparison of Femtosecond Laser Assisted Cataract Surgery to Conventional Phacoemulsification Cataract Surgery on Corneal Endothelial Cell Loss
Brief Title: Comparison of Femtosecond Laser Assisted Cataract Surgery to Conventional Phacoemulsification Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00089916
Record Dates: First submitted 2014-03-16; First posted 2014-03-26 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Cataract
Keywords: Cataract, femtosecond laser, FLACS
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- conventional: Patients who undergo routine cataract surgery using conventional phacoemulsification technique
- FLACS: Patients who undergo femtosecond laser assisted cataract surgery

SUMMARY:
In this project, the investigators aim to compare the safety, efficacy, and predictability outcomes of conventional CEIOL surgery to Femtosecond-laser-assisted CEIOL (FLACS) in an effort to improve cataract surgery outcomes. The investigators hypothesis is that FLACS may lead to preservation of endothelial cells compared to conventional CE IOL.

DETAILED DESCRIPTION:
This study will only include patients who are eligible to undergo cataract surgery. All patients will receive treatment that is FDA approved for cataract surgery. Because all study participants will have been scheduled for elective cataract extraction regardless of their participation in this study, there will be little or no additional surgical risk associated with participation. A total of 720 patients are expected to be enrolled in the study during a period of 2 years. The investigators will recruit patients with bilateral operable cataracts. One eye will undergo cataract surgery using conventional cataract extraction technique including phacoemulsification whereas the second eye will undergo FLACS. No significant increased risk to the patient is expected in either arm of the study compared to routine cataract surgery. The patients will be examined as per previous post-operative cataract surgery guidelines on POD1, POW1, POM1, POM3, POM6, POY1 and POY2. The only treatment difference will take place at the time of the cataract surgery. Post-operatively, endothelial cell count will be obtained by the no-touch technology of specular microscopy at baseline as well as three months after surgery. If the study ends prematurely, the investigators do not anticipate any significant change in the care of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years of age
2. Ability to understand and sign an informed consent
3. Visually significant cataract eligible to undergo cataract extraction by phacoemulsification with primary intraocular lens implantation in at least 1 eye
4. Ability and commitment to follow up for 18 months after surgery
5. No other ocular pathology and no previous/concurrent surgery

Exclusion Criteria:

1. Any other ocular pathology that may affect best-corrected visual acuity
2. Previous or concurrent ocular surgery
3. Subjects who are pregnant, lactating, or planning to be pregnant during the course of the study.
4. Patients with keratoconus or keratectasia
5. Patients who are blind on one eye

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to our center with visually significant cataract and who may benefit from cataract surgery
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2014-05; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
endothelial cell density three months after conventional CEIOL or FLACS compared to baseline | up to 2 years
  endothelial cell density will be compared at baseline and three months after a patient undergoes FLACS or Conventional CE IOL to see which technique causes less endothelial cell loss.

CONTACTS AND LOCATIONS:
Overall Officials: yassine daoud, md, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States